CLINICAL TRIAL: NCT04710758
Title: Prospective Randomized Controlled Multicenter Clinical Trial For Comparison Of Long-term Outcomes Between Laparoscopic And Open Total Gastrectomy In Patients With Locally Advanced Gastric Cancer
Brief Title: Multicenter Study on Laparoscopic Total Gastrectomy for Advanced Gastric Cancer
Acronym: CLASS-07
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-006
Record Dates: First submitted 2021-01-02; First posted 2021-01-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Laparoscopic total gastrectomy; Open total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic total gastrectomy (Experimental): The surgeon will perform LTG with D2 lymphadenectomy for patients enrolled in this group.
  Interventions: Procedure: Laparoscopic total gastrectomy
- Open total gastrectomy (Active Comparator): The surgeon will perform OTG with D2 lymphadenectomy for patients enrolled in this group.
  Interventions: Procedure: Open total gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic total gastrectomy — LTG with D2 lymphadenectomy for patients with locally advanced gastric cancer (clinical stage T2-4aN0-3M0)
  Other Names: Experimental group (LTG)
  Arms: Laparoscopic total gastrectomy
Procedure: Open total gastrectomy — OTG with D2 lymphadenectomy for patients with locally advanced gastric cancer (clinical stage T2-4aN0-3M0)
  Other Names: Control group (OTG)
  Arms: Open total gastrectomy

SUMMARY:
CLASS-07 trial is a prospective, multicenter, randomized controlled trial for comparison of long-term outcomes between laparoscopic total gastrectomy (LTG) and open total gastrectomy (OTG) in patients with locally advanced gastric cancer (clinical stage T2-4aN0-3M0). The primary purpose of this study is to evaluate the overall survival and determine the efficacy of LTG compared with OTG for locally advanced gastric cancer. The second purpose is to evaluate the 3-year overall survival rate, 3-year disease free survival rate, morbidity and mortality rates, 3-year recurrence pattern and postoperative recovery course of the patients enrolled in this study.

DETAILED DESCRIPTION:
Gastric cancer is a significant global health problem, especially in East Asia. With an increase in the incidences of proximal gastric cancer over the last decades, the value of total gastrectomy is more emphasized. Laparoscopic total gastrectomy (LTG) has become an attracting option for surgeons due to its well-known advantages. However, more evidence is needed to support the safety and efficacy of LTG in locally advanced gastric cancer.

Recently，a multicenter, open-label, noninferiority, randomized clinical trial (CLASS-02) launched by Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group compared the safety of LTG for clinical stage I gastric cancer with open total gastrectomy (OTG). The overall morbidity and mortality rates were 19.1% in the LTG group and 20.2% in the OTG group, which was not significantly different (rate difference, -1.1%). This study demonstrated that LTG can be safely performed by experienced surgeons for clinical stage I gastric cancer. However, there hasn't been any prospective randomized clinical trial study evaluating the safety and efficacy of LTG in advanced gastric cancer.

This CLASS-07 trial is a prospective, multicenter, randomized controlled trial for comparison of long-term outcomes between LTG and OTG in patients with locally advanced gastric cancer (clinical stage T2-4aN0-3M0). The primary purpose of this study is to evaluate the overall survival and determine the efficacy of LTG compared with OTG for locally advanced gastric cancer. The second purpose is to evaluate the 3-year overall survival rate, 3-year disease free survival rate, morbidity and mortality rates, 3-year recurrence pattern and postoperative recovery course of the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years
2. Tumor located in the middle or upper third of the stomach, and curative resection is expected to be achievable by total gastrectomy with D2 lymphadenectomy (also apply to multiple primary cancers);
3. Primary lesion is pathologically diagnosed as gastric adenocarcinoma, such as papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly cohesive carcinoma (including signet ring cell carcinoma and other variants), and mixed adenocarcinoma;
4. Clinical stage T2-4aN0-3M0 (According to AJCC-8th TNM staging system);
5. Expected survival > 6 months
6. No invasion to Z-line;
7. BMI (Body Mass Index) < 30 kg/m2
8. No history of upper abdominal surgery (except for laparoscopic cholecystectomy);
9. No prior treatment of chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc
10. Preoperative performance status (ECOG，Eastern Cooperative Oncology Group) of 0 or 1
11. Preoperative ASA (American Society of Anesthesiologists) scoring: I-III
12. Sufficient organ functions
13. Written informed consent

Exclusion Criteria:

1. Preoperative examinations indicate regional fusion of enlarged lymph nodes (max diameter ≥ 3.0cm) or enlargment of spleen hilus lymph nodes
2. Women during pregnancy or breast-feeding
3. Synchronous or metachronous (within 5 years) malignancies
4. Body temperature ≥ 38℃ before surgery or infectious disease with a systemic therapy indicated
5. Severe mental disease
6. Severe respiratory disease, FEV1 < 50% of predicted
7. Severe hepatic and renal dysfunction
8. Unstable angina pectoris or history of myocardial infarction within 6 months
9. History of cerebral infarction or cerebral hemorrhage within 6 months
10. Continuous systemic steroid therapy within 1 month (except for topical use)
11. Gastric cancer complications (bleeding, perforation, obstruction) that requiring emergency surgery
12. Patients are participating or have participated in another clinical trial (within 6 months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1018 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Overall survival (OS) was defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
3-year overall survival rate | 3 years
  # of patients who are still alive at 3 years out of all study patients
3-year disease free survival rate | 3 years
  # of patients who are free of gastric cancer at 3 years out of all study patients
Early morbidity rate | 30 days
  The early morbidity are defined as the event observed within 30 days following surgery, including intraoperative and postoperative complications
Early mortality rate | 30 days
  The early mortality are defined as the event observed within 30 days following surgery, including intraoperative and postoperative death
3-year recurrence pattern | 3 years
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Postoperative recovery course | 30 days
  Time to first ambulation, flatus, liquid diet, and soft diet are used to assess the postoperative recovery course, which is a composite outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Yihong Sun, MD, Principal Investigator — Fudan University
Locations (1):
- ZhongShan hospital FuDan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Yang L, Zheng R, Wang N, Yuan Y, Liu S, Li H, Zhang S, Zeng H, Chen W. Incidence and mortality of stomach cancer in China, 2014. Chin J Cancer Res. 2018 Jun;30(3):291-298. doi: 10.21147/j.issn.1000-9604.2018.03.01. PMID 30046223
- [Background] Yamashita H, Seto Y, Sano T, Makuuchi H, Ando N, Sasako M; Japanese Gastric Cancer Association and the Japan Esophageal Society. Results of a nation-wide retrospective study of lymphadenectomy for esophagogastric junction carcinoma. Gastric Cancer. 2017 Mar;20(Suppl 1):69-83. doi: 10.1007/s10120-016-0663-8. Epub 2016 Oct 28. PMID 27796514
- [Background] Liu K, Yang K, Zhang W, Chen X, Chen X, Zhang B, Chen Z, Chen J, Zhao Y, Zhou Z, Chen L, Hu J. Changes of Esophagogastric Junctional Adenocarcinoma and Gastroesophageal Reflux Disease Among Surgical Patients During 1988-2012: A Single-institution, High-volume Experience in China. Ann Surg. 2016 Jan;263(1):88-95. doi: 10.1097/SLA.0000000000001148. PMID 25647058
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Background] Katai H, Mizusawa J, Katayama H, Takagi M, Yoshikawa T, Fukagawa T, Terashima M, Misawa K, Teshima S, Koeda K, Nunobe S, Fukushima N, Yasuda T, Asao Y, Fujiwara Y, Sasako M. Short-term surgical outcomes from a phase III study of laparoscopy-assisted versus open distal gastrectomy with nodal dissection for clinical stage IA/IB gastric cancer: Japan Clinical Oncology Group Study JCOG0912. Gastric Cancer. 2017 Jul;20(4):699-708. doi: 10.1007/s10120-016-0646-9. Epub 2016 Oct 7. PMID 27718137
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2018 (5th edition). Gastric Cancer. 2021 Jan;24(1):1-21. doi: 10.1007/s10120-020-01042-y. Epub 2020 Feb 14. No abstract available. PMID 32060757
- [Background] Lee HJ, Hyung WJ, Yang HK, Han SU, Park YK, An JY, Kim W, Kim HI, Kim HH, Ryu SW, Hur H, Kong SH, Cho GS, Kim JJ, Park DJ, Ryu KW, Kim YW, Kim JW, Lee JH, Kim MC; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Short-term Outcomes of a Multicenter Randomized Controlled Trial Comparing Laparoscopic Distal Gastrectomy With D2 Lymphadenectomy to Open Distal Gastrectomy for Locally Advanced Gastric Cancer (KLASS-02-RCT). Ann Surg. 2019 Dec;270(6):983-991. doi: 10.1097/SLA.0000000000003217. PMID 30829698
- [Background] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Background] Yu J, Huang C, Sun Y, Su X, Cao H, Hu J, Wang K, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Hu Y, Liu H, Zheng C, Li P, Xie J, Liu F, Li Z, Zhao G, Yang K, Liu C, Li H, Chen P, Ji J, Li G; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Effect of Laparoscopic vs Open Distal Gastrectomy on 3-Year Disease-Free Survival in Patients With Locally Advanced Gastric Cancer: The CLASS-01 Randomized Clinical Trial. JAMA. 2019 May 28;321(20):1983-1992. doi: 10.1001/jama.2019.5359. PMID 31135850
- [Background] Kawamura H, Yokota R, Homma S, Kondo Y. Comparison of invasiveness between laparoscopy-assisted total gastrectomy and open total gastrectomy. World J Surg. 2009 Nov;33(11):2389-95. doi: 10.1007/s00268-009-0208-y. PMID 19760315
- [Background] Wang W, Zhang X, Shen C, Zhi X, Wang B, Xu Z. Laparoscopic versus open total gastrectomy for gastric cancer: an updated meta-analysis. PLoS One. 2014 Feb 18;9(2):e88753. doi: 10.1371/journal.pone.0088753. eCollection 2014. PMID 24558421
- [Background] Hyung WJ, Yang HK, Han SU, Lee YJ, Park JM, Kim JJ, Kwon OK, Kong SH, Kim HI, Lee HJ, Kim W, Ryu SW, Jin SH, Oh SJ, Ryu KW, Kim MC, Ahn HS, Park YK, Kim YH, Hwang SH, Kim JW, Cho GS. A feasibility study of laparoscopic total gastrectomy for clinical stage I gastric cancer: a prospective multi-center phase II clinical trial, KLASS 03. Gastric Cancer. 2019 Jan;22(1):214-222. doi: 10.1007/s10120-018-0864-4. Epub 2018 Aug 20. PMID 30128720
- [Background] Katai H, Mizusawa J, Katayama H, Kunisaki C, Sakuramoto S, Inaki N, Kinoshita T, Iwasaki Y, Misawa K, Takiguchi N, Kaji M, Okitsu H, Yoshikawa T, Terashima M; Stomach Cancer Study Group of Japan Clinical Oncology Group. Single-arm confirmatory trial of laparoscopy-assisted total or proximal gastrectomy with nodal dissection for clinical stage I gastric cancer: Japan Clinical Oncology Group study JCOG1401. Gastric Cancer. 2019 Sep;22(5):999-1008. doi: 10.1007/s10120-019-00929-9. Epub 2019 Feb 20. PMID 30788750
- [Background] He H, Li H, Su X, Li Z, Yu P, Huang H, Huang C, Ye J, Li Y, Suo J, Yu J, Li G, Xu Z, Zhao G, Cao H, Hu J, Du X, Liu F, Sun Y; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Study on safety of laparoscopic total gastrectomy for clinical stage I gastric cancer: the protocol of the CLASS02-01 multicenter randomized controlled clinical trial. BMC Cancer. 2018 Oct 3;18(1):944. doi: 10.1186/s12885-018-4846-z. PMID 30285673
- [Background] Liu F, Huang C, Xu Z, Su X, Zhao G, Ye J, Du X, Huang H, Hu J, Li G, Yu P, Li Y, Suo J, Zhao N, Zhang W, Li H, He H, Sun Y; Chinese Laparoscopic Gastrointestinal Surgery Study (CLASS) Group. Morbidity and Mortality of Laparoscopic vs Open Total Gastrectomy for Clinical Stage I Gastric Cancer: The CLASS02 Multicenter Randomized Clinical Trial. JAMA Oncol. 2020 Oct 1;6(10):1590-1597. doi: 10.1001/jamaoncol.2020.3152. PMID 32815991